CLINICAL TRIAL: NCT05607069
Title: Multifactorial Evaluation of COVID-19 Respiratory Reliquates
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Sponsor
Other Study IDs: 00097/2022
Record Dates: First submitted 2022-11-04; First posted 2022-11-07 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: COVID-19 Respiratory Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 previous infection

SUMMARY:
The present study aims to evaluate how commonly diagnostic tools employed in the preoperative evaluation of respiratory function in thoracic surgery can identify pathological alteration due to a previous SARS-CoV-2 infection. In particular, the investigators will gather information concerning imaging (lung ct and lung ultrasound), arterial blood gas analysis, and pulmonary function tests.

ELIGIBILITY:
Inclusion Criteria:

* previous SARS-Cov2 infection
* awaiting lung resection surgery

Exclusion Criteria:

* less than 18 years of age
* unable to consent to enroll
* refuse to enroll

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll patients scheduled for lung resection surgery that had a documented previous SARS-Cov2 infection.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-05-28 (Actual); Primary Completion 2023-05-28 (Actual); Study Completion 2024-05-28 (Estimated)

PRIMARY OUTCOMES:
sensibility of preoperative evaluation in identifying pathological sequelae due to SARS-Cov2 infection | 12 month

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Città della Salute e della Scienza di Torino, Turin, Italy

IPD SHARING:
Plan to Share IPD: No